CLINICAL TRIAL: NCT02578316
Title: An Open-Label, Non-Randomized, Single-Center Study to Determine the Metabolism and Elimination of 14C-E7080 in Patients With Advanced Solid Tumors or Lymphomas, Who Are Unsuitable For, or Have Failed, Existing Therapies.
Brief Title: A Study to Determine the Metabolism and Elimination of 14C-E7080 in Patients With Advanced Solid Tumors or Lymphomas, Who Are Unsuitable For, or Have Failed, Existing Therapies.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-E044-104
Record Dates: First submitted 2015-10-15; First posted 2015-10-16 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-04

CONDITIONS: Advanced Solid Tumors; Lymphomas
Keywords: Advanced Solid Tumors; Lymphomas
MeSH Terms: conditions — Lymphoma | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenvatinib 24 mg (Experimental): Participants with advanced solid tumors or lymphomas, who are unsuitable for, or had failed, existing therapies.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Study phase dosing: participants received an initial single dose of radiolabelled 14C-lenvatinib oral patient dosing solution containing 24 mg of lenvatinib as anhydrous free base and radioactivity of 3.7 millibecquerel (MBq) on Day 1.
  Extension phase dosing: 24 mg of 14C-lenvatinib: 2 x 10mg, and 4 x 1mg or 1 x 4mg tablets once-daily, continuously in each 28-day cycle during extension phase.
  Other Names: E7080, Lenvima

SUMMARY:
The purpose of this study was to determine the metabolism and elimination of 14C-lenvatinib in participants with advanced solid tumors or lymphomas, who were unsuitable for, or had failed, existing therapies.

DETAILED DESCRIPTION:
The study comprised of two phases, the Study Phase and Extension Phase. Participants received 14C-lenvatinib on Day 1 of the Study Phase. Thereafter participants were given daily oral doses of 24 mg of lenvatinib over a 28 day cycle. During the Study Phase, participants received an initial single dose of 14C-lenvatinib oral patient dosing solution containing 24 mg of lenvatinib as anhydrous free base and radioactivity of 100 mCi (3.7 MBq) on Day 1, followed by collection of blood, urine and feces samples for pharmacokinetic analysis between Day 1 and Day 8, with a discharge visit on Day 8. Participants then entered the Extension Phase of the study to continue to receive once daily oral administration of non-radiolabeled lenvatinib at a dose of 24 mg. Each 28-day dosing period will be considered one treatment cycle.

ELIGIBILITY:
INCLUSION CRITERIA

1. Participants with histologically and/or cytologically confirmed solid tumor or lymphoma who were resistant/ refractory to approved therapies or for whom no appropriate therapies were available. Participants with measurable tumors according to RECIST were desirable but not essential for inclusion.
2. All previous treatment (including surgery and radiotherapy) must have been completed at least four weeks prior to study entry and any acute toxicity must have resolved
3. Aged greater than or equal to 18 years
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
5. Could take oral study medication
6. Gave written informed consent to participate in the study
7. Willing and complied with the study protocol for the duration of the study.

EXCLUSION CRITERIA

1. Participants with brain or subdural metastases, unless they had completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs and/or symptoms of brain metastases those were stable for at least 4 weeks.
2. Participants with meningeal carcinomatosis
3. Any of the following values for laboratory parameters:

   1. hemoglobin less than 9 g/dL (5.6 mmol/L);
   2. neutrophils less than 1.5 x 10^9/L;
   3. platelets less than 100 x 10^9/L;
   4. Prothrombin time (PT) [or International Normalized Ratio (INR)] and Patial thromboplastin time (PTT) > 1.5 x the upper limit of normal (ULN)
   5. serum bilirubin greater than 1.5 x ULN
   6. other liver parameters greater than 3 x ULN
   7. creatinine clearance less than 60 mL/min per the Cockcroft and Gault formula
4. Uncontrolled infections
5. Significant cardiovascular impairment (history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable ischemic heart disease including a myocardial infarction within six months of study start, or serious cardiac arrhythmia)
6. Participants with marked baseline prolongation of QT/QT interval corrected for heart rate (QTc) interval (QTc interval greater than or equal to 500 msec) using the Fridericia method
7. Any treatment with an investigational drug within the last 30 days
8. Women who were pregnant or breast-feeding; women of childbearing potential with a positive pregnancy test at screening or no pregnancy test. Women of child-bearing potential unless (1) surgically sterile or (2) using adequate measures of contraception in the opinion of the Investigator (including two forms of contraception, one of which must be a barrier method). Perimenopausal women who were amenorrheic for at least 12 months to be considered of non-child-bearing potential. Fertile males with female partners of child-bearing potential who were not willing to use contraception, or whose female partners were not using adequate contraceptive protection, were excluded.
9. Proteinuria greater than 1+ on bedside testing
10. History of gastrointestinal malabsorption
11. Surgery within four weeks of start of study treatment
12. Bleeding or thrombotic disorders or use of an anticoagulant, such as warfarin, with a therapeutic INR. Aspirin, non-steroidal anti-inflammatory drugs (NSAIDs), and low molecular weight heparin (LMWH) were permissible but when used with caution.
13. Poorly controlled hypertension (defined as a change in hypertensive therapy within three months of study start) or participants diagnosed with hypertension (defined as a repeat blood pressure measurement of 160/90 mmHg or higher) at screening
14. Previous lenvatinib therapy
15. History of alcoholism, drug addiction, psychiatric or psychological condition, or social situation which, in the opinion of the investigator, would impair study compliance
16. History of allergic reactions attributed to compounds of similar chemical or biological composition to lenvatinib
17. Other significant disease or disorder that, in the Investigator's opinion, would exclude the participant from the study
18. Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam, Netherlands

REFERENCES:
- [Background] Dubbelman AC, Rosing H, Mejui-Roelvink M, Gupta A, Verbel D, Sellecchia R, et al. A mass balance study of 14C-lenvatinib (E7080) in patients with advanced solid tumours or lymphomas. Presented at the Scientific Meeting of the Dutch Society for Clinical Pharmacology and Biopharmacy (NVKFB); 2012 Mar 30; Utrecht (The Netherlands). 2012. Dubbelman AC, Rosing H, Thijssen B, Gebretensae A, Lucas L, Chen H, et al. Development and validation of LC-MS/MS assays for the quantification of E7080 and metabolites in various human biological matrices. J Chromatogr B, 2012; 887-888:25-34.

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenvatinib: Study Phase: Participants received a single dose of an oral dosing solution of 14^C-labeled lenvatinib (approximately 100 μCi or 3.7 MBq) and approximately 24 mg non-radiolabeled lenvatinib on Day 1. From Days 1 to 8, participants remained in the research unit so blood, urine, and fecal samples could be collected for PK analysis and determination of 14^C-lenvatinib concentrations prior to, and for 7 days following, drug administration. Participants were discharged after the checkout procedures were completed on Day 8, or when the level of radiation in urine and fecal samples was less than 1% of the total radioactive dose.
  Extension Phase: Participants received 24 mg oral lenvatinib once daily at home or at the clinic on Visit Days 1, 8, 15, and 22 of each treatment cycle (1 treatment cycle = 28 days) until discontinuation from the study. The dose of lenvatinib could be reduced or discontinued during any cycle because of toxicity
Period: Study Phase
Arm/Group | Lenvatinib
Started | 6
Completed | 6
Not Completed | 0
Period: Extension Phase
Arm/Group | Lenvatinib
Started | 6
Completed | 0
Not Completed | 6
Not completed — Progression of disease | 6

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least a partial dose of study drug and had at least one postdose safety assessment.
Groups:
- Lenvatinib: Study Phase: Participants received a single dose of an oral dosing solution of 14^C-labeled lenvatinib (approximately 100 μCi or 3.7 MBq) and approximately 24 mg non-radiolabeled lenvatinib on Day 1. From Days 1 to 8, participants remained in the research unit so blood, urine, and fecal samples could be collected for pharmacokinetic (PK) analysis and determination of 14^C-lenvatinib concentrations prior to, and for 7 days following, drug administration. Participants were discharged after the checkout procedures were completed on Day 8, or when the level of radiation in urine and fecal samples was less than 1% of the total radioactive dose.
  Extension Phase: Participants received 24 mg oral lenvatinib once daily at home or at the clinic on Visit Days 1, 8, 15, and 22 of each treatment cycle (1 treatment cycle = 28 days) until discontinuation from the study. The dose of lenvatinib could be reduced or discontinued during any cycle because of toxicity.
Arm/Group | Lenvatinib
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.8 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Radiolabeled 14^C-Lenvatinib and Non-Radiolabeled Lenvatinib
Description: Blood samples were drawn at specific time points then analyzed for the amount of 14^C-lenvatinib and non-radiolabeled lenvatinib in the plasma. Individual blood/plasma concentration-time data were analyzed using 'non-compartmental' analysis. Cmax was determined from visual inspection of the individual blood/plasma concentration-time profile and was summarized as the Geometric Mean and percent coefficient of variation for the Geometric Mean (CV%) for all participants and expressed as nanograms/milliliter (ng/mL).
Time Frame: Day 1 (pre-dose, post-dose at 15 and 30 minutes, 1, 2, 4, 6, 8 and 12 hours), Day 2 (24 hours), Day 3 (48 hours), Day 4 (72 hours), Day 5 (96 hours), Day 6 (120 hours), Day 7 (144 hours) and Day 8 (168 hours)
Population: The Pharmacokinetic (PK) Analysis Set is the group of participants who received the Study Phase dose of 14^C-lenvatinib and have any evaluable post 14^C- lenvatinib dose plasma and/or blood concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 14^C-Lenvatinib: Study Phase: Participants received a single dose of an oral dosing solution of 14^C-labeled lenvatinib (approximately 100 μCi or 3.7 MBq) and approximately 24 mg non-radiolabeled lenvatinib on Day 1. From Days 1 to 8, participants remained in the research unit so blood, urine, and fecal samples could be collected for PK analysis and determination of 14^C-lenvatinib concentrations prior to, and for 7 days following, drug administration. Participants were discharged after the checkout procedures were completed on Day 8, or when the level of radiation in urine and fecal samples was less than 1% of the total radioactive dose.
  Extension Phase: Participants received 24 mg oral lenvatinib once daily at home or at the clinic on Visit Days 1, 8, 15, and 22 of each treatment cycle (1 treatment cycle = 28 days) until discontinuation from the study. The dose of lenvatinib could be reduced or discontinued during any cycle because of toxicity.
Arm/Group | 14^C-Lenvatinib | Lenvatinib
Number analyzed (Participants) | 6 | 6
ng/mL | 485.2 (37.08) | 426.8 (46.59)

2. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of Radiolabeled 14^C-Lenvatinib and Non-Radiolabeled Lenvatinib
Description: Blood samples were drawn at specific time points then analyzed for the amount of 14^C-lenvatinib and non-radiolabeled lenvatinib in the plasma. Individual blood/plasma concentration-time data were analyzed using 'non-compartmental' analysis. Tmax was determined from visual inspection of the individual blood/plasma concentration-time profile and was summarized as the Geometric Mean (CV%) for all participants and expressed as hours.
Time Frame: as for outcome 1
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 14^C-Lenvatinib | Lenvatinib
Number analyzed (Participants) | 6 | 6
Hours | 1.418 (41.95) | 1.604 (39.33)

3. Primary Outcome: Terminal Phase Rate Constant (λz) of Radiolabeled 14^C-Lenvatinib and Non-Radiolabeled Lenvatinib in Plasma
Description: Blood samples were drawn at specific time points then analyzed for the amount of 14^C-lenvatinib and non-radiolabeled lenvatinib in the plasma. The terminal phase rate constant represents the rate at which study drug was eliminated from the body and was determined by log-linear regression of the plasma concentrations against time in the terminal phase and was summarized as the Geometric Mean (CV%) for all participants and expressed as 1/hours.
Time Frame: as for outcome 1
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | 14^C-Lenvatinib | Lenvatinib
Number analyzed (Participants) | 6 | 6
1/hour | 0.039 (39.5787) | 0.020 (24.7258)

4. Primary Outcome: Terminal Exponential Half-life (t1/2) of Radiolabeled 14^C-Lenvatinib and Non-Radiolabeled Lenvatinib in Plasma
Description: Blood samples were drawn at specific time points then analyzed for the amount of 14^C-lenvatinib and non-radiolabeled lenvatinib in the plasma. The terminal phase t1/2 is the time required to divide the plasma concentration of study drug by two after reaching pseudo-equilibrium, and not the time required to eliminate half of the administered dose of study drug. The t1/2 during the apparent terminal disposition phase was calculated at 0.693/λz and was summarized as the Geometric Mean (CV%) for all participants and expressed as hours.
Time Frame: as for outcome 1
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 14^C-Lenvatinib | Lenvatinib
Number analyzed (Participants) | 6 | 6
Hours | 17.78 (39.44) | 34.54 (25.12)

5. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Time t (AUC(0-t))
Description: Blood samples were drawn at specific time points then analyzed for the amount of 14^C-lenvatinib and non-radiolabeled lenvatinib in the plasma. The AUC(0-t) was calculated by the combination of linear/log (from Tmax) trapezoidal rule where 't' is the time of last quantifiable plasma concentration following dosing. AUC(0-t) was summarized as the Geometric Mean (CV%) for all participants and expressed in nanograms·hour/milliliter (ng·hr/mL).
Time Frame: as for outcome 1
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Arm/Group | 14^C-Lenvatinib | Lenvatinib
Number analyzed (Participants) | 6 | 6
ng·hr/mL | 5223 (55.00) | 3440 (49.72)

6. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC(0-inf))
Description: Blood samples were drawn at specific time points then analyzed for the amount of 14^C-lenvatinib and non-radiolabeled lenvatinib in the plasma. The AUC(0-inf) was calculated as AUC(0-t) + Ct/λz where Ct is the last measurable concentration and was summarized as the Geometric Mean (CV%) for all participants and expressed in ng·hr/mL.
Time Frame: as for outcome 1
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Arm/Group | 14^C-Lenvatinib | Lenvatinib
Number analyzed (Participants) | 6 | 6
ng·hr/mL | 5783 (48.22) | 3469 (49.95)

7. Primary Outcome: Percentage of Area Under the Plasma Concentration Curve Extrapolated to Infinity (%AUC(Extra))
Description: Blood samples were drawn at specific time points then analyzed for the amount of 14^C-lenvatinib and non-radiolabeled lenvatinib in the plasma. %AUC(extra) was calculated as [(AUC(0-inf) - AUC(0-t)/AUC(0-inf) ]*100 and was summarized as the Geometric Mean (CV%) for all participants and expressed in (ng·hr/mL).
Time Frame: as for outcome 1
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent lenvatinib
Arm/Group | 14^C-Lenvatinib | Lenvatinib
Number analyzed (Participants) | 6 | 6
Percent lenvatinib | 8.637 (46.9657) | 0.786 (44.2610)

8. Primary Outcome: Apparent Clearance (CL/F) of Lenvatinib From Plasma
Description: Blood samples were drawn at specific time points then analyzed for the amount of 14^C-lenvatinib and non-radiolabeled lenvatinib in the plasma. The CL/F for parent lenvatinib only was calculated as Dose/[AUC(0-inf)] and was summarized as the Geometric Mean (CV%) for all participants and expressed in L/hr.
Time Frame: as for outcome 1
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | Lenvatinib
Number analyzed (Participants) | 6
L/hour | 6.739 (49.54)

9. Primary Outcome: Apparent Terminal Volume of Distribution in the Terminal Phase of Lenvatinib (Vz/F)
Description: Blood samples were drawn at specific time points then analyzed for the amount of 14^C-lenvatinib and non-radiolabeled lenvatinib in the plasma. Vz/F for lenvatinib only was calculated as Dose/[(λz)·(AUC(0-inf))] and was summarized as the Geometric Mean (CV%) for all participants and expressed in liters (L).
Time Frame: as for outcome 1
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Lenvatinib
Number analyzed (Participants) | 6
L | 335.7 (36.69)

10. Primary Outcome: Renal Clearance of Lenvatinib (CLr)
Description: CLr was determined based on the interval amount and cumulative amount of the analyte excreted in the urine divided by its corresponding AUC over the same collection interval. Aeurine(0-t)/AUC(0-t), where t is the last measurable concentration, was calculated for lenvatinib only and was summarized as the Geometric Mean (CV%) for all participants and expressed in L/hr.
Time Frame: Pre-dose, post-dose at 0-6, 6-12, 12-18, 18-24, 24-30, 30-36, 36-42, 42-48, 48-72, 72-96, 96-120, 120-144, and 144-168 hours
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | Lenvatinib
Number analyzed (Participants) | 6
L/hour | 0.042 (140.3)

11. Primary Outcome: Percentage Recovery of 14^C- Lenvatinib Related Material in the Urine
Description: Urine samples were collected at specific time points, then analyzed for the amount of 14^C- lenvatinib related material. The total radioactive dose of 14^C-lenvatinib excreted in urine (Aeurine%) was calculated from the time of dosing to the last quantifiable measurement. If radioactivity levels were still present at the end of the Study Phase, sampling continued until each sample contained less than 1% of the total radioactive dose. Percentage recovery of 14^C- lenvatinib related material in the urine was summarized as the Geometric Mean (CV%) percent cumulative for all participants and expressed as percent of 14^C- lenvatinib.
Time Frame: as for outcome 10
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of 14^C-lenvatinib
Arm/Group | 14^C-Lenvatinib
Number analyzed (Participants) | 6
Percentage of 14^C-lenvatinib | 24.74 (17.76)

12. Primary Outcome: Percentage Recovery of 14^C- Lenvatinib Related Material in the Feces
Description: Fecal samples were collected at specific time points, then analyzed for the amount of 14^C- lenvatinib related material. The percentage of the 14^C- lenvatinib dose excreted in feces (Aefeces%) was calculated from time of dosing to the last quantifiable measurement. If radioactivity levels were still present at the end of the Study Phase, sampling continued until each sample contained less than 1% of the total radioactive dose. Percentage recovery of 14^C- lenvatinib related material in the feces was summarized as the Geometric Mean (CV%) percent cumulative for all participants and expressed as percent of 14^C- lenvatinib.
Time Frame: Day 1 to Day 8
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of 14^C-lenvatinib
Arm/Group | 14^C-Lenvatinib
Number analyzed (Participants) | 6
Percentage of 14^C-lenvatinib | 63.56 (11.24)

13. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Safety was assessed by monitoring and recording all AEs including all Common Terminology Criteria for Adverse Events (CTCAE) grades (for both increasing and decreasing severity) and SAEs; regular monitoring of hematology, blood chemistry, and urine values; results of physical examinations, regular measurement of vital sign measurements, and 12-lead electrocardiogram (ECG), as detailed in the Schedule of Visits and Procedures. The relationship of AEs to treatment was based on investigator judgment. Details of AEs and SAEs are provided in the reported adverse event section.
Time Frame: Date of first dose of study treatment till 30 days after the last dose, assessed up to 1 year
Population: The Safety Analysis Set was the group of participants who received at least one partial dose of study drug and had at least one postdose safety assessment.
Measure: Number; unit: Percentage of participants
Groups:
- 14C^Lenvatinib/Lenvatinib: Study Phase: Participants received a single dose of an oral dosing solution of 14^C-labeled lenvatinib (approximately 100 μCi or 3.7 MBq) and approximately 24 mg non-radiolabeled lenvatinib on Day 1. From Days 1 to 8, participants remained in the research unit so blood, urine, and fecal samples could be collected for PK analysis and determination of 14^C-lenvatinib concentrations prior to, and for 7 days following, drug administration. Participants were discharged after the checkout procedures were completed on Day 8, or when the level of radiation in urine and fecal samples was less than 1% of the total radioactive dose.
  Extension Phase: Participants received 24 mg oral lenvatinib once daily at home or at the clinic on Visit Days 1, 8, 15, and 22 of each treatment cycle (1 treatment cycle = 28 days) until discontinuation from the study. The dose of lenvatinib could be reduced or discontinued during any cycle because of toxicity.
Arm/Group | 14C^Lenvatinib/Lenvatinib
Number analyzed (Participants) | 6
Percentage of participants
  Any TEAEs | 100
  Treatment-related TEAEs | 100
  Serious TEAEs | 50.0
  TEAEs requiring study drug reduction | 33.3
  TEAEs requiring dose interruption | 83.3

14. Secondary Outcome: Objective Tumor Response
Description: A response of complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) was assigned by the investigator as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0. CR was defined as disappearance of all target lesions. Any pathological lymph node had to be reduced in short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameter. PD was defined as a 20% or greater increase in the sum of the longest diameter of measured lesions, taking as reference the smallest sum longest diameter recorded since treatment start or the appearance of one or more new lesions. CR or PR was confirmed no less than 4 weeks after first observation of the response. For SD, measurements must have met the SD criteria at least once after study entry at a minimum interval of 6 weeks. SD is defined as lasting at least 5 weeks.
Time Frame: Baseline to first date of documented CR, PR, SD, or PD, assessed up to 1 year
Population: The Response Evaluable Population is the group of participants who received at least a partial dose of study treatment who had measureable disease per RECIST at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | 14C^Lenvatinib/Lenvatinib
Number analyzed (Participants) | 6
Percentage of participants
  Complete response | 0
  Partial Response | 16.7
  Stable disease | 50.0
  Progressive disease | 33.3

ADVERSE EVENTS:
Time Frame: Approximately 17 months.
Description: Treatment-emergent adverse events (TEAEs) were defined as any event with start date/time beyond or equal to the day of initial dosing, and/or any adverse event (AE) for which an increase in severity occurs during the trial. All AEs were graded according to National Cancer Institute Common Toxicity Criteria for Adverse Events version 3.0.
Arm/Group | Lenvatinib
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib (N=6)
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib (N=6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Glossodynia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Disease progression (General disorders) | 2
Fatigue (General disorders) | 4
Feeling cold (General disorders) | 2
Oedema peripheral (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Cystitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Blood pressure increased (Investigations) | 1
Weight decreased (Investigations) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4
Blister (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No